CLINICAL TRIAL: NCT00464633
Title: A Multicenter, Open-label, Single Arm Study of Weekly Alvocidib in Patients With Previously Treated B-Cell Chronic Lymphocytic Leukemia (CLL) or Prolymphocytic Leukemia (PLL) Arising From CLL
Brief Title: Alvocidib in Patients With Previously Treated Chronic Lymphocytic Leukemia or Prolymphocytic Leukemia Arising From Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC6663; 2006-006152-34 (EudraCT Number)
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Leukemia, Lymphocytic, Chronic
Keywords: CLL; PLL; flavopiridol
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — alvocidib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alvocidib (Experimental): Cycles with 4-week treatment with alvocidib followed by 2-week rest period for up to a maximum of 6 cycles
  Interventions: Drug: alvocidib

INTERVENTIONS:
Drug: alvocidib — 1st dose: 30 mg/m2 as a 30-minute intravenous (IV) infusion followed by 30 mg/m2 as a 4-hour continuous infusion
  Then, every treatment week, depending upon the patient's objective response to initial therapy:
  * 30 mg/m2 over 30 minutes followed by 50 mg/m2 over 4 hours or
  * 30 mg/m2 over 30 minutes followed by 30 mg/m2 over 4 hours.
  Other Names: HMR1275

SUMMARY:
Multicenter, open-label, study of alvocidib in previously treated chronic lymphocytic leukemia patients.

Primary objective is to determine overall response rate.

The secondary objectives are:

* to assess overall safety,
* to assess duration of response, progression free survival, and overall survival.

Clinical benefit and pharmacokinetics parameters are also evaluated.

DETAILED DESCRIPTION:
Treatment until disease progression or no evidence of treatment response; occurrence of unacceptable toxicity, intercurrent medical problem, or adverse event (AE); or a maximum of 6 cycles.

Follow-up of 6 months after the last treatment with alvocidib.

The maximum duration of the study participation for patient will be about 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have documentation of histologically confirmed and measurable Chronic Lymphocytic Leukemia (CLL) or Prolymphocytic Leukemia (PLL) arising from CLL;
* Patient must have symptomatic and progressive disease;
* Patient must have received prior alkylating agent(s) and be fludarabine refractory;
* Patient must have the adequate organ functions;
* Patient's Eastern Cooperative Oncology Group performance (ECOG) status must be 0-2;

Exclusion Criteria:

* Patient with de novo PLL;
* Patient with secondary malignancy that will limit survival ≤5 years;
* Patient with prior allogenic or autologous bone marrow transplant or peripheral blood stem cell transplant ≤12 months;
* Patient receiving an investigational agent or an approved agent for an investigational purpose within last 4 weeks prior to study entry;
* Patient with known history of glucose-6-phosphate dehydrogenase deficiency;
* Patient with autoimmune hemolytic anemia;
* Patient with known Central Nervous System involvement;
* Patient with active, uncontrolled serious bacterial, viral or fungal infections

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2007-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Best overall objective response rate | Up to a maximum of 6 cycles
  Objective Response Rate (ORR) is defined as the proportion of participants with complete response or partial response (including nodular partial response) relative to the total number of participants.
  Response assessment is based on evaluation of nodal disease by Computerized Tomography (CT) and National Cancer Institute Working Group 96 criteria (NCI-96) for assessment of liver, spleen, constitutional symptoms, peripheral blood (±) bone marrow.

SECONDARY OUTCOMES:
Progression-free survival | Up to a maximum of 6 cycles
  Progression-free survival (PFS) is defined as the time from the date of first administration of study drug to the first documentation of progressive disease or death due to any cause in the absence of previous documentation of objective progression.
Duration of objective response | Up to a maximum of 6 cycles
  Duration of objective response is defined from the time of first occurrence of complete response or partial response (including nodular partial response) to the first documentation of progressive disease or death due to any cause in the absence of previous documentation of objective progression.
Overall survival | Up to a maximum of 6 cycles
  Overall survival (OS) is defined as the time from the date of first administration of study drug to death.
Overview of adverse events | from study drug administration up to 30 days after last study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (34):
- United States (13):
  - Sanofi-Aventis Investigational Site Number 840008, San Diego, California
  - Sanofi-Aventis Investigational Site Number 840022, San Francisco, California
  - Sanofi-Aventis Investigational Site Number 840010, Chicago, Illinois
  - Sanofi-Aventis Investigational Site Number 840012, Chicago, Illinois
  - Sanofi-Aventis Investigational Site Number 840017, Indianapolis, Indiana
  - Sanofi-Aventis Investigational Site Number 840001, Boston, Massachusetts
  - Sanofi-Aventis Investigational Site Number 840023, Ann Arbor, Michigan
  - Sanofi-Aventis Investigational Site Number 840005, New York, New York
  - Sanofi-Aventis Investigational Site Number 840006, New York, New York
  - Sanofi-Aventis Investigational Site Number 840003, Durham, North Carolina
  - Sanofi-Aventis Investigational Site Number 840018, Cleveland, Ohio
  - Sanofi-Aventis Investigational Site Number 840002, Columbus, Ohio
  - Sanofi-Aventis Investigational Site Number 840020, Philadelphia, Pennsylvania
- Sanofi-Aventis Investigational Site Number 036001, St Leonards, Australia
- Belgium (5):
  - Sanofi-Aventis Investigational Site Number 056006, Bruges
  - Sanofi-Aventis Investigational Site Number 056001, Brussels
  - Sanofi-Aventis Investigational Site Number 056004, Ghent
  - Sanofi-Aventis Investigational Site Number 056003, Leuven
  - Sanofi-Aventis Investigational Site Number 056002, Yvoir
- France (3):
  - Sanofi-Aventis Investigational Site Number 250001, Paris
  - Sanofi-Aventis Investigational Site Number 250003, Pierre-Bénite
  - Sanofi-Aventis Investigational Site Number 250002, Tours
- Germany (3):
  - Sanofi-Aventis Investigational Site Number 276001, Cologne
  - Sanofi-Aventis Investigational Site Number 276004, Kiel
  - Sanofi-Aventis Investigational Site Number 276002, Ulm
- Italy (2):
  - Sanofi-Aventis Investigational Site Number 380002, Bologna
  - Sanofi-Aventis Investigational Site Number 380001, Milan
- Netherlands (3):
  - Sanofi-Aventis Investigational Site Number 528003, Amsterdam
  - Sanofi-Aventis Investigational Site Number 528001, Groningen
  - Sanofi-Aventis Investigational Site Number 528002, Rotterdam
- Sanofi-Aventis Investigational Site Number 630001, San Juan, Puerto Rico
- United Kingdom (3):
  - Sanofi-Aventis Investigational Site Number 826005, Aberdeen
  - Sanofi-Aventis Investigational Site Number 826002, Birmingham
  - Sanofi-Aventis Investigational Site Number 826004, Bournemouth